CLINICAL TRIAL: NCT01593540
Title: Clinical Efficacy and Patient Acceptance of Metal and Metal-Free Interdental Brushes: A Controlled Prospective Randomized Study
Brief Title: Clinical Examination of Metal Free Interdental Brushes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Johan Wölber, DDS, Principal investigator, Dr., University of Freiburg
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: woel-01
Record Dates: First submitted 2012-04-28; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Gingivitis; Periodontitis
MeSH Terms: conditions — Gingivitis; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- metal-free interdental brushes. (Experimental)
  Interventions: Device: metal-free interdental brush
- metal-core interdental brushes (Active Comparator)
  Interventions: Device: metal-core interdental brush

INTERVENTIONS:
Device: metal-free interdental brush — one time per day
  Other Names: Fuchs brush&clean
  Arms: metal-free interdental brushes.
Device: metal-core interdental brush — one time per day
  Other Names: TePe Interdental brushes
  Arms: metal-core interdental brushes

SUMMARY:
The aim of the study was to evaluate the clinical efficacy (Eastman Interdental Bleeding Index, Quigley and Hein) of a novel metal-free interdentalbrush compared to a classig metal-core interdental brush.

DETAILED DESCRIPTION:
Self-performed interdental cleaning is a crucial element in preventing gingival or periodontal diseases. Interdental cleaning is most efficiently performed through usage of interdental brushes. Commonly used metal-core interdental brushes can harbour the risk of hard tissue damage when used inappropriately.The aim of the study was to evaluate the clinical efficacy and patient satisfaction of a novel metal-free interdental brush. This was tested on healthy participants. The control group performed interdental cleaning with a commonly used metal-core interdental brush.

ELIGIBILITY:
Inclusion Criteria:

* minimum age: 18 years

Exclusion Criteria:

* allergy against one or more parts of the interdental brushes
* non-treated periodontitis
* soft-tissue changes of the mucosa
* orthodontic treatment
* removable prosthesis
* pregnancy
* anticoagulants
* drugs causing gingivahyperplasia
* indications for antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Analysis of the differences between both groups. Measurements in form of Plaque-Index (Quigley und Hein, Tureskey Mod. 1970) | Beginning and after four weeks of use

SECONDARY OUTCOMES:
Eastman Interdental Bleeding Index, questionnaire of patient acceptance | Beginning and after four weeks of use

CONTACTS AND LOCATIONS:
Overall Officials: Johan P Woelber, Dr., Study Director — University of Freiburg
Locations (1):
- University Freiburg Medical Center , Dept of Operative Dentistry and Periodontology, Freiburg im Breisgau, Germany